CLINICAL TRIAL: NCT05514912
Title: Optimal Preoperative Therapy for Intrahepatic Cholangiocarcinoma (OPTIC)
Brief Title: Preoperative Nab-paclitaxel, Cisplatin, and Gemcitabine Chemotherapy With or Without Infigratinib Targeted Therapy for the Treatment of Resectable Intrahepatic Cholangiocarcinoma, The OPTIC Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI has decided to terminate this study due to study supporter pulling support on this study.
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shishir Kumar Maithel, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004206; NCI-2022-05975 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00004206 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5569-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Resectable Intrahepatic Cholangiocarcinoma; Stage 0 Intrahepatic Cholangiocarcinoma AJCC v8; Stage I Intrahepatic Cholangiocarcinoma AJCC v8; Stage II Intrahepatic Cholangiocarcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; infigratinib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (nab-paclitaxel, cisplatin, gemcitabine, infigratinib) (Experimental): While awaiting NGS molecular profile results, all patients receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8 of one 21-day cycle in the absence of disease progression or unacceptable toxicity.
  Patients who are FGFR2 fusion/translocation positive receive infigratinib PO QD for days 1-21 of each cycle. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients whose cancer is stable or improved undergo surgery to remove the tumor within 8 weeks of completing preoperative therapy per standard of care.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Drug: Infigratinib Phosphate; Drug: Nab-paclitaxel
- Arm B (nab-paclitaxel, cisplatin, gemcitabine) (Active Comparator): While awaiting NGS molecular profile results, all patients receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8 of one 21-day cycle in the absence of disease progression or unacceptable toxicity.
  Patients who are FGFR2 fusion/translocation negative continue receiving nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients whose cancer is stable or improved undergo surgery to remove the tumor within 8 weeks of completing preoperative therapy per standard of care.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Drug: Infigratinib Phosphate — Given PO
  Other Names: N'-(2,6-Dichloro-3,5-dimethoxyphenyl)-N-(6-(4-(4-ethylpiperazin-1-yl)anilino)pyrimidin-4-yl)-N-methylurea Phosphate (1:1); Truseltiq
  Arms: Arm A (nab-paclitaxel, cisplatin, gemcitabine, infigratinib)
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel

SUMMARY:
This phase II trial assesses the feasibility (including both safety and tolerability) of conducting Next Generation Sequencing and administering targeted therapy (infigratinib) in the preoperative setting for patients with intrahepatic cholangiocarcinoma that can be removed by surgery (resectable). Chemotherapy drugs, such as nab-paclitaxel, cisplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Targeted therapy with infigratinib will bind to FGFR which can help stop tumor cell growth and cause tumor cell death. Giving chemotherapy and/or targeted therapy before surgery may make the tumor smaller for resection and may help prevent the cancer from coming back. If a molecular profiling test shows a genetic change called an FGFR2 fusion, patients receive both chemotherapy and targeted therapy while patients without a FGFR2 fusion just receive chemotherapy. Giving targeted therapy based on molecular profile testing results prior to attempted resection of an intrahepatic cholangiocarcinoma that has a risk for either not being able to be removed or for coming back after it has been removed may help improve treatment outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of a novel treatment strategy that includes conducting next generation sequencing (NGS)-based treatment on a preoperative tissue biopsy and subsequent administration of infigratinib phosphate (infigratinib) to patients with FGFR2 fusions versus neoadjuvant chemotherapy consisting of gemcitabine hydrochloride (gemcitabine), cisplatin, and nab-paclitaxel to all other patients for resectable intrahepatic cholangiocarcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the intervention by assessing the radiological response rate.

II. To assess degree of pathologic response in the surgical specimen. III. To assess response to therapy by measuring circulating tumor deoxyribonucleic acid (CT-DNA).

IV. To determine the R0 resection rate. V. To determine recurrence-free survival (RFS). VI. To determine overall survival (OS).

OUTLINE:

While awaiting NGS molecular profile results, all patients receive nab-paclitaxel intravenously (IV) over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8 of one 21-day cycle in the absence of disease progression or unacceptable toxicity.

After obtaining NGS molecular profile results, patients who are FGFR2 fusion/translocation positive are assigned to Arm A, while patients who are FGFR2 fusion/translocation negative are assigned to Arm B.

ARM A: Patients receive infigratinib orally (PO) once daily (QD) on days 1-21 of each cycle. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients whose cancer is stable or improved undergo surgery to remove the tumor within 8 weeks of completing preoperative therapy per standard of care.

ARM B: Patients continue receiving nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients whose cancer is stable or improved undergo surgery to remove the tumor within 8 weeks of completing preoperative therapy per standard of care.

After completion of study treatment, patients are followed up within 4 weeks and every 4 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intrahepatic cholangiocarcinoma
* High-quality cross-sectional imaging by computerized tomography (CT) or magnetic resonant imaging (MRI) performed within 6 weeks prior to enrollment and showed a resectable IHCCA confined to the liver, bile duct, and /or regional lymph nodes. No distant extrahepatic disease is allowed.
* Adults > 18 years of age
* Able to give informed consent
* Able to adhere to study visit schedule and other protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate bone marrow reserves as evidenced by:
* Absolute neutrophil count (ANC) ≥1,500 cells/ul
* Platelet count ≥100,000 cells/μl
* Hemoglobin ≥9 g/dL
* Adequate hepatic function as evidenced by:
* Serum total bilirubin ≤1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN
* Albumin ≥3 g/dl
* Adequate renal function as evidenced by creatinine ≤1.5 x ULN
* Creatinine =< 1.5 x ULN
* Have amylase or lipase < 2.0 x ULN
* Male, or a non-pregnant and non-lactating female
* Women of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must commit to true abstinence from heterosexual contact, or agree to use, and be able to comply with, effective contraception without interruption for 28 days prior to starting gemcitabine/cisplatin/nab- paclitaxel (including dose interruptions) until treatment with gemcitabine/cisplatin/nab-paclitaxel is complete.
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a female of childbearing potential or a pregnant female while on treatment (including during dose interruptions) with gemcitabine/cisplatin/nab-paclitaxel and for 6 months following gemcitabine/cisplatin/nab- paclitaxel is continuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0. In CTCAE version 4.0 grade 2 sensory neuropathy is defined as "moderate symptoms; limiting instrumental activities of daily living (ADLs)".
* Have current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, inflammation or ulceration, keratoconjunctivitis, confirmed by ophthalmic examination. Subjects with asymptomatic ophthalmic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study.
* Have used medications known to prolong the QT interval and/or are associated with a risk of Torsades de Pointes (TdP) 7 days prior to first dose of study drug.
* Have consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products containing juice of these fruits within 7 days prior to first dose of study drug.
* Have current evidence of concerning endocrine alterations of calcium/phosphate homeostasis, eg, parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc, in the opinion of the investigator.
* Have abnormal calcium or phosphorus, or calcium-phosphorus product ≥55 mg^2 /dL2:

  * Inorganic phosphorus above local normal limits
  * Total corrected serum calcium above local normal limits
* Are currently receiving or are planning to receive during participation in this study, treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs.
* Have clinically significant cardiac disease including any of the following: a. Congestive heart failure requiring treatment (New York Heart Association Grade ≥2), or uncontrolled hypertension (refer to the European Society of Cardiology and European Society of Hypertension guidelines (Williams et al 2018)
* Fridericia's correction formula QTcF >470 msec (males and females). Note: If the QTcF is >470 msec in the first ECG, a total of 3 ECGs separated by at least 5 minutes should be performed. If the average of these 3 consecutive results for QTcF is ≤470 msec, the subject meets eligibility in this regard
* Known history of congenital long QT syndrome
* Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, symptomatic congestive heart failure, uncontrolled diabetes, serious active, uncontrolled infection after inadequate biliary drainage if tumor obstructing bile duct, or psychiatric illness/social situations.
* Pregnancy (positive pregnancy test) or lactation.
* Known CNS disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Previous (within the past 3 years) or concurrent presence of other cancer, except non-melanoma skin cancer, renal cell carcinoma < 3cm, neuroendocrine tumors < 2cm, and in situ carcinomas including bronchoalveolar carcinoma (BAC).
* History of allergy or hypersensitivity to any of the study drugs.
* Current abuse of alcohol or illicit drugs.
* Inability or unwillingness to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Completing All Preoperative Testing and Therapy | Up to 3 years
  Treatment completion is defined as completion of next generation sequencing testing and all preoperative and operative therapy. The completion of all therapy rate, along with the exact 95% binomial confidence interval will be record. If a patient is not a candidate for surgery after completion of all preoperative therapy, this will be considered an event against feasibility of this treatment strategy, at which time patients will receive further treatment as best deemed by their treating physician.
Unacceptable Toxicity | Up to 3 years
  Unacceptable toxicity is defined as any grade 3 or higher toxicities by Common Terminology Criteria for Adverse Events criteria that result in a treatment delay of >4 weeks. The rate of unacceptable toxicity will be reported, along with the exact 95% binomial confidence interval. If the therapy cannot be completed due to a delay of >4 weeks, this will be considered an event for this approach not being feasible.
Safety and Tolerability | Up to 3 years
  Safety and tolerability will be assessed in terms of adverse events, and serious adverse events. Summary of these events will be tabulated by the maximum reported Common Terminology Criteria for Adverse Events grade and in relation to study treatment. Both adverse Events and serious adverse events will be tabulated using frequencies and percentages.

SECONDARY OUTCOMES:
Radiological Response Rate by Response Evaluation Criteria in Solid Tumors | Up to 3 years
  Radiological response rate will be defined as the percentage of patients who will have complete response, partial response or stable disease after the neoadjuvant therapy. The radiological response rate will be estimated, along with the exact 95% binomial confidence interval.
Pathologic Response Rate | Up to 3 years
  Pathologic response will be defined as the degree of treatment effect to preoperative therapy. This will be measured as percent of viable cancer cells and percent of necrotic cells in the surgically resected specimen. A pathologic complete response is defined as having no viable cancer cells in the surgical specimen at the time of surgery.
Circulating Tumor Deoxyribonucleic Acid Response | Up to 3 years
  Circulating tumor deoxyribonucleic acid will be collected as an exploratory secondary endpoint. The investigators will be blinded as to the results of the circulating tumor deoxyribonucleic acid assay until after the study is complete as to avoid any bias towards treatment decisions based on this exploratory endpoint.
Recurrence-Free Survival | Time between the date of surgery and the date of disease recurrence or death, whichever occurred first, or assessed up to 3 years
  Recurrence-free survival is defined as the time between the date of surgery and the date of disease recurrence or death, whichever occurred first. If a patient did not have an event (i.e. disease recurrence or death) by the time of final analysis, patient will be censored at the last disease evaluation time. The Kaplan-Meier method will be used to estimate recurrence-free survival. The two-sided log-rank tests will be used to assess the differences of recurrence-free survival between groups.
Overall Survival | Time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive, or assessed up to 3 years
  Overall survival is defined as the time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date. The Kaplan-Meier method will be used to estimate overall survival. The two-sided log-rank tests will be used to assess the differences of overall survival between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shishir K. Maithel, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute